CLINICAL TRIAL: NCT05079308
Title: Clinical Trial on the Level of Respiratory Protection of Surgical Face Masks and Filtering Face Pieces (FFP2), With and Without a Peripheral Sealing Device, Against Covid-19
Brief Title: Clinical Trial on the Efficacy of Different Masks With and Without a Peripheral Sealing Device, Against Covid-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: UBalearicIslands
Record Dates: First submitted 2021-09-08; First posted 2021-10-15 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Covid19; Personal Protective Equipment
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Filtering face piece with peripheral sealing device (Experimental): Individuals using the Filtering face Piece (FFP2) with the Peripheral Sealing Device (AMS).
  Interventions: Device: Peripheral sealing device for surgical mask or filtering face piece
- Filtering face piece without peripheral sealing device (Active Comparator): Individuals using the Filtering face Piece (FFP2) without the AMS;
  Interventions: Device: Peripheral sealing device for surgical mask or filtering face piece
- IIR surgical mask with peripheral sealing device (Experimental): Individuals using the Surgical mask (SM) with the AMS;
  Interventions: Device: Peripheral sealing device for surgical mask or filtering face piece
- IIR surgical mask without peripheral sealing device (Active Comparator): Individuals using the Surgical mask (SM) without the AMS;
  Interventions: Device: Peripheral sealing device for surgical mask or filtering face piece
- Filtering face piece with IIR surgical mask (Experimental): individuals using a FFP2 with a SM over it, simultaneously, without the AMS.
  Interventions: Device: IIR Surgical mask with Filtering face piece

INTERVENTIONS:
Device: Peripheral sealing device for surgical mask or filtering face piece — The individuals used a Peripheral Sealing Device on a surgical mask or a filtering face piece mask and were submitted to a qualitative fit test, regulated by the Occupational Security and Health Administration (USA).
  Arms: Filtering face piece with peripheral sealing device; Filtering face piece without peripheral sealing device; IIR surgical mask with peripheral sealing device; IIR surgical mask without peripheral sealing device
Device: IIR Surgical mask with Filtering face piece — The individuals used a IIR surgical mask with a filtering face piece mask and were submitted to a qualitative fit test, regulated by the Occupational Security and Health Administration (USA).
  Arms: Filtering face piece with IIR surgical mask

SUMMARY:
A significant number of professionals subjected to high-risk situations have been infected by Covid-19, due to the lack of adequate respiratory protection equipment or poor marginal sealing adjustments. Then, the objective of this study is to determine if there are statistically significant differences in the level of respiratory protection of type IIR surgical face masks and filtering face masks, used with and without a peripheral sealing device, against the contagion of Covid-19 or other harmful biological agents. The proposed device is a thermoplastic resin ring composed of a reusable and biodegradable polylactic acid designed to be used in a healthcare environment. The individuals of the study will be submitted to qualitative fit tests, that meet current Ocupational Security and Health Administration (OSHA) standard. The mentioned qualitative fit test uses a sodium saccharin solution to evaluate the respiratory protection equipment in professionals in hospitals, emergency centers, and early childhood education centers.

DETAILED DESCRIPTION:
The purpose of the research is to determine if there are statistically significant differences in the level of respiratory protection in situations of high risk against the contagion of Covid-19 or other harmful biological agents, in subjects who use filtering face pieces (FFP2) with or without a peripheral sealing device (AMS), Type IIR surgical face masks with or without a AMS, and subjects using the FFP2 filtering face mask simultaneously with the Type IIR surgical face mask. For this, a total of 210 individuals were selected from different environments in order to attain diversity, while controlling for representativeness bias. They were selected from the ADEMA University School - UIB, nursing staff from the Infectious Diseases Service at Son Espases University Hospital, 112 Emergency Service of the Autonomous Community of the Balearic Islands and the General Directorate of Planning and Centers of the Ministry of Education and Professional Training (Balearic Islands, Spain).

Participants were assigned to one of the 5 groups and subgroups, after accepting their participation in the study voluntarily and freely by signing the consent form approved by the CEI-IB.

To evaluate the adjustment of the respiratory protective equipment with and without the personalized peripheral sealing device (AMS), a sweet sensitivity test was performed with the 3M FT-10 Qualitative Fit-Test Kit (Saint Paul, Minnesota, USA), which complies with the current standards of the Occupational Security and Health Administration (OSHA) and according to the protocol described in Riutord-Sbert et al. (2021). During the qualitative fit test, a total of seven mobility exercises of 60 seconds each were performed, and the nebulizer was squeezed, every 30 seconds:

Phase 1 - Normal breathing Phase 2 - Slow and deep breathing Phase 3 - Breathing whilst moving the head to both sides Phase 4 - Breathing whilst moving the head up and down Phase 5 - Breathing spelling the alphabet Phase 6 - Breathing whilst moving up and down from the waist Phase 7 - Normal breathing

If the fit test was completed within 7 minutes without the individual having detected the sweet taste, the seal was considered optimal or adequate and the experiment was graded as APPROVED. If the subject detected the sweet test before seven minutes, the adjustment was considered inadequate and was scored as FAILED, noting the time it took to detect the sweet taste as established in the protocol of the 3M FT-10 Fit test (Riutord-Sbert et al. 2021).

ELIGIBILITY:
Inclusion Criteria:

* people familiar with the use of face masks, absence of allergy or intolerance to sodium saccharin or materials used, absence of relevant systemic diseases, age between 18-65 years, absence of obvious facial hair and signing the informed consent.

Exclusion Criteria:

* people not familiar with the use of face masks, presence of allergy or intolerance to sodium saccharin or materials used, presence of relevant systemic diseases, presence of obvious facial hair and not signing the informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis of the respiratory protective equipment in protecting against the simulated aerosol: intergroup comparison | up to 5 months
  A qualitative analysis will be performed in order to evaluate whether the respiratory protective equipment is effective in protecting the individuals from a simulated aerosol environment. The individuals will be submitted to 7 different breathing exercises inside of a hood with their open mouth. A nebulizer filled with sacharin solution will be used to simulate an aerosol environment. If the individual do not sense the taste during the whole breathing exercises (total of 7 minutes) the respiratory protective equipment (RPE) used by this individual will be scored as "PASSED". If the individial sense the sweet taste during the 7 minutes, the RPE will be scored as "FAILED". The answer of the individuals using masks with the Peripheral Sealing Device and the controls (individual using masks without the peripheral sealing device) within each group will be compared. There is only one outcome measure: evaluate if the individuals are able to sense the aeresol or not.

SECONDARY OUTCOMES:
Qualitative analysis of the respiratory protective equipment in protecting against the simulated aerosol: intragroup comparison | up to 5 months
  A qualitative analysis will be performed in order to evaluate whether the respiratory protective equipment (RPE) tested in the study are effective in protecting the individuals from a simulated aerosol environment. Subjects of the Subgroup FFP2 with AMS with the subjects of the Subgroup SM with AMS; the subjects of the Subgroup FFP2 with AMS with those of the subjects of the Group FFP2+SM and, finally, the subjects of the SM with AMS with the subjects of the FFP2+SM Group. There is only one outcome measure: evaluate if the individuals are able to sense the aeresol or not.

CONTACTS AND LOCATIONS:
Locations (1):
- ADEMA University School, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: No